CLINICAL TRIAL: NCT03432234
Title: Respiratory Microbiome and COPD Exacerbations
Brief Title: Respiratory Microbiome and COPD Exacerbations (RESMECOPD)
Acronym: RESMECOPD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Corporacion Parc Tauli (Other)
Collaborators: Hospital de Sant Pau (Other); Hospital Clinic of Barcelona (Other); Hospital Universitari de Bellvitge (Other); Hospital del Mar (Other); Germans Trias i Pujol Hospital (Other); Hospital Arnau de Vilanova (Other); Centre for Genomic Regulation (Unknown)
Responsible Party: Principal Investigator, Eduard Monsó-Molas, Head of Respiratory Medicine Department, Corporacion Parc Tauli
Other Study IDs: PI15/0157 (2015607)
Record Dates: First submitted 2018-01-08; First posted 2018-02-14 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Exacerbation COPD
Keywords: COPD; Microbiome; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Biomarkers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Oral Wash, oropharingeal swab, sputum, brochoalveolar lavage, feces, plasma, serum, white blood cells.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD and frequent exacerbation: Patient with COPD diagnosis and at least two exacerbations by year (FE)
  Interventions: Other: Biomarkers
- COPD no frequent exacerbation: Patient with COPD diagnosis with no frequent exacerbation, less than 2 by year (NE).
  Interventions: Other: Biomarkers
- Healthy (control): Healthy volunteers patients (H)
  Interventions: Other: Biomarkers

INTERVENTIONS:
Other: Biomarkers — This is an observational study, there is no intervention

SUMMARY:
The global objective of this coordinated project is to test the following hypotheses: 1) the lung microbiome in chronic obstructive pulmonary disease (COPD) is different in patients suffering from frequent exacerbations (FE) compared those who do not (NE ); 2) The microbial profile of patients with FE is associated with a different local and systemic inflammatory pattern; and 3) the inflammatory and immune characteristics of COPD are modulated by the intestinal microbiome.

The project is based on bronchoalveolar lavage (BAL) for sampling lung microbiome, and includes analysis of regional variability (intrapulmonary) and temporal variability. The project will also assess the correlation between BAL samples obtained from the proximal airway (oral cavity, oropharynx and sputum), and the representation of lung microbiome in them. A cohort of COPD patients (n = 50 FE; n = 50 NE) and healthy subjects (n= 30), matched by age, sex and tobacco consumption. Respiratory secretion samples will be collected in clinical stability samples, with resampling in a quarter of the participants at 6-9 months. Coordinator Project: Bacterial and fungal microbiota will be determined by 16S rRNA and ITS amplification and sequencing. Virome and functional metagenomics will be analyzed in a quarter of the participants. Subprojects: Regional variability in the lung, local and systemic inflammatory response, and the relationship between the intestinal microbiome and inflammatory and clinical characteristics of the disease will be determined. The integration of the results will be performed using network medicine methodologies. The results of this project will help to understand the pathogenesis of COPD and its exacerbations with the final aim to identify new therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Spirometry: FEV1/FVC < 70%; FEV1 between 50 and 80% predicted (GOLD II/III)
* Clinical Stability (no therapeutic change and/or use of antibiotics) during 8 weeks. - The treatment received will be registered for post-hoc studies stratified by this condition.

Exclusion Criteria:

* Drug addiction, alcohol abuse,
* Use of long-term oral or nebulised antibiotic therapy.
* History of allergies, asthma or other chronic respiratory disease, sanitary worker, working exposure to dust or fumes.
* Other diseases: Severe cardiovascular, neurological, psychiatric, renal, hepatic or gastrointestinal , that might interfere with the daily life activities.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible subjects were COPD patients GOLD II/III in stable situation.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-03-07 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Respiratory Microbiome in COPD patients with FE and NE. | 7 days
  Respiratory Microbiome composition will be determined by using metagenomic aproaches.

SECONDARY OUTCOMES:
Bacteria related to pulmonary and systemic inflamatory factors (FE vs NE) | 7 days
  Determination of pulmonary and systemic markers with ELISA kit. Microbiome will be determined by metagenomic techniques.
Longitudinal variability of respiratory microbiome in COPD patients (FE vs NE). | 12 months
  Change of respiratory Microbiome (diversity and abundance)
Inmunological response of lung epithelial cells COPD patients after an infectious and inflammatory stimuli | 7 days
  The in vitro response of epithelial cells will be determined with ELISA kits.

OTHER OUTCOMES:
Spatial variability of respiratory microbiome in COPD patients (FE vs NE). | 1 day
  Respiratory Microbiome Composition of different types of samples.

CONTACTS AND LOCATIONS:
Overall Officials: Oriol Sibila, Principal Investigator — Hospital de Sant Pau; Rosa Faner, Principal Investigator — Hospital Clínic; Eduard Monso, Study Director — Hospital Parc Tauli
Locations (6):
- Spain (6):
  - Corporació Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic, Barcelona
  - Hospital de Bellitge, Barcelona
  - Hospital del Mar, Barcelona
  - Hosptial de Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
Sequencing data will be available in public databases.